CLINICAL TRIAL: NCT02351297
Title: Effects of High Protein Diet on the Large Intestine in Overweight Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Avicenne (Other)
Responsible Party: Principal Investigator, Robert Benamouzig, Head of gastroenterology department, Hospital Avicenne
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2013-A01730-45
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Overweight; Healthy
Keywords: High protein diet; Microbiota; Rectal biopsies; Metabolomics; Bacterial metabolites; volunteers
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Casein supplementation (Experimental): After the run-in period, volunteers will receive casein supplementation (15 % of energy intake) for 3 weeks.
  Interventions: Dietary Supplement: casein supplementation
- Soy protein supplementation (Experimental): After the run-in period, volunteers will receive soy protein supplementation (15 % of energy intake) for 3 weeks.
  Interventions: Dietary Supplement: soy protein supplementation
- Maltrodextrin supplementation (Placebo Comparator): After the run-in period, volunteers will receive maltodextrin supplementation (15 % of energy intake) for 3 weeks.
  Interventions: Dietary Supplement: maltodextrin supplementation

INTERVENTIONS:
Dietary Supplement: casein supplementation — After the run-in period, volunteers will receive casein supplementation (15 % of energy intake) for 3 weeks.
  Arms: Casein supplementation
Dietary Supplement: soy protein supplementation — After the run-in period, volunteers will receive soy protein supplementation (15 % of energy intake) for 3 weeks.
  Arms: Soy protein supplementation
Dietary Supplement: maltodextrin supplementation — After the run-in period, volunteers will receive maltodextrin supplementation (15 % of energy intake) for 3 weeks.
  Arms: Maltrodextrin supplementation

SUMMARY:
This study aims at evaluating the consequences of a 3 weeks high protein diet on the large intestine ecosystem (microbiota, metabolites and gene expression in rectal mucosa). Those parameters will be analysed with technics including OMICs methods. After a run-in period, 42 volunteers will receive either soy or milk protein or maltodextrin as a placebo control. This trial is double blind randomized placebo-controlled paralleled design (3 arms). Longitudinal sampling will allow the comparison of parameters during the study.

DETAILED DESCRIPTION:
High protein diets are widely used for their slimming effect. Those diets increase the quantity of undigested protein and peptides reaching the large intestine. Microbiota utilizes protein and peptides as substrates and produces amino-acid derived metabolites such as short chain fatty acids, branched chain fatty acids, lactate, formate, succinate, ammonium, hydrogen sulfide and phenolic compounds. Some of those metabolites have been shown to be beneficial to the host whereas other could be deleterious. High protein diets may have different effects whether based on animal or plant proteins since those two kinds of protein have different amino acids composition and slightly different digestibility. The objective of this study is to evaluate in overweight volunteers the consequences of high protein diets (animal vs vegetal) vs isocaloric-normoproteic diet at the level of the large intestine and metabolism. Firstly, composition and activity of the microbiota and the metabolites produced in the large intestine lumen will be determined. Then, to evaluate the consequences of the tested diets on mucosal physiology, gene expression will be analyzed in rectal biopsies and fecal water will be tested on colonocytes cell lines. Lastly, the consequences of the diets on host metabolism will be evaluated.

Dietary intervention

Before the study, volunteers (n=42) will provide a 3 day food record that will be utilized by a dietician to calculate their usual energy intake. The study will start with a 2 weeks normalization period during which the volunteers will have to eat according to menus (Fig. 1). The diet will provide to the volunteer their usual individual energy intake; and protein, carbohydrates and fat will respectively provide 15, 50 and 35 % of the energy intake.

At the end of this standardization period, volunteers will be randomly assigned into 3 groups (n=14) for 3 weeks (intervention period) (Fig. 1). Volunteers of the 3 groups will follow a diet with a reduced digestible carbohydrates intake (15% of energy intake) while undigestible carbohydrate intake will remain unchanged. The volunteers will consume 3 times per day a dietary supplement powder that they will dissolve in water and then drink. This supplement will provide them 15% of their energy intake. The first group will receive a casein (animal protein) supplement so that they will have a high protein diet (protein, carbohydrates and fat will respectively provide 30, 35 and 35 % of the energy intake). The second group will receive a soy protein(vegetal) supplement so that they will also consume a high protein diet (protein, carbohydrates and fat will respectively provide 30, 35 and 35 % of the energy intake). The third group will receive a maltodextrin (digestible carbohydrate, placebo control) supplement so that they will ingest a normoproteic diet, similar in macronutrient composition to the standardization diet (protein, carbohydrates and fat will respectively provide 15, 50 and 35 % of the energy intake). The dietary supplement will be given in a double-blinded protocol. There will be no energy restriction between the standaridization and intervention periods.

Clinical protocol

Daily, the volunteers will measure their body weight and record their food consumption and physical activity. Once a week, they will have a phone call with a dietician to ensure dietary compliance (Fig. 2).

At the end of the normalization period, 13 days after the beginning of the study (D13), volunteers will collect 24h urine samples. Stool samples will be collected from the evening of D13 to the morning of D14 . A cooler will be provided to the volunteer for storage and transport of samples. After one night fasting, in the morning of D14, the volunteers will come to the hospital and will bring their samples that will be immediately conditioned for storage. Blood samples will be collected. Then, rectal biopsies will be recovered. Every week during the intervention period, urine stool and blood will be sampled (D21, D28, D35). At the end of the intervention period, rectal biopsies will be recovered (D35). Body weight and blood pressure will be measured at each visit.

Analyses All measured parameters will be expressed relatively to baseline.

Dietary intake will be evaluated by dietician based on food records.

Stool samples

* Microbiota composition and functions
* Luminal metabolites composition
* pH, osmolarity, water content
* Fecal water test on HT-29 cells (colonocytes) for mitochondrial respiration, proliferation, genotoxicity, cytotoxicity, gene expression

Urines

* Urea and creatinine assay (protein consumption marker to verify dietary compliance)
* Metabolomics

Blood

* Clinical parameters (total cholesterol, LDL and HDL cholesterol, non-esterified fatty acids, triglycerides, glycemia, insulinemia)
* Metabolomics

Rectal biopsies

• Transcriptomic analyses

ELIGIBILITY:
Inclusion Criteria:

* BMI 25- 30
* Body weight stable last 3 months
* Moderate physical activity

Exclusion Criteria:

* Abnormal food behavior
* Digestive, renal, hepatic, pulmonary, hemostasis, neoplasic diseases
* antibiotic, pre or probiotics use in the last 3 months
* intolerance for the tested product
* positive serology for infectious disease
* pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in gene expression in rectal biopsy from baseline after 3 week dietary intervention | Change for baseline in gene expression in rectal biopsy after 3 weeks dietary intervention
  Gene expression in biopsies collected before (baseline) and after 3 week dietary intervention will be measured by transcriptomic analyses. Differential gene expression will be expressed as relative units (fold change).

SECONDARY OUTCOMES:
microbiota composition analysis | Change for baseline in microbiota composition after 3 weeks dietary intervention
  Microbiota composition will be analysed in stool samples before (baseline) and after 3 week dietary intervention using metagenomic analyses and will be expressed as bacterial relative abundance.
fecal water metabolomics | Change for baseline in fecal water metabolites after 3 weeks dietary intervention
  Fecal water metabolites will be analysed in stool samples before (baseline) and after 3 week dietary intervention using RMN analyses and will be expressed as metabolites relative abundance.

CONTACTS AND LOCATIONS:
Overall Officials: Robert BENAMOUZIG, MD PhD, Principal Investigator — Avicenne Hospital

REFERENCES:
- [Derived] Beaumont M, Portune KJ, Steuer N, Lan A, Cerrudo V, Audebert M, Dumont F, Mancano G, Khodorova N, Andriamihaja M, Airinei G, Tome D, Benamouzig R, Davila AM, Claus SP, Sanz Y, Blachier F. Quantity and source of dietary protein influence metabolite production by gut microbiota and rectal mucosa gene expression: a randomized, parallel, double-blind trial in overweight humans. Am J Clin Nutr. 2017 Oct;106(4):1005-1019. doi: 10.3945/ajcn.117.158816. Epub 2017 Sep 13. PMID 28903954